CLINICAL TRIAL: NCT02360397
Title: Ranolazine Mediated Premature Ventricular Contraction Reduction in Ischemic Heart Disease
Brief Title: Ranolazine Mediated PVC Reduction in Ischemic Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kent Hospital, Rhode Island (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Chester Hedgepeth, MD, PhD, Chester Hedgepeth, MD, PhD, Kent Hospital, Rhode Island
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-259-1341
Record Dates: First submitted 2015-01-20; First posted 2015-02-10 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Ventricular Premature Complexes; Myocardial Ischemia
MeSH Terms: conditions — Ventricular Premature Complexes; Myocardial Ischemia | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranolazine (Experimental): Ranolazine 1000 mg tablet twice daily for 30 days
  Interventions: Drug: ranolazine

INTERVENTIONS:
Drug: ranolazine — Ranolazine 1000 mg tablet twice daily for 30 days
  Other Names: ranexa

SUMMARY:
The purpose of this study is to determine whether ranolazine has beneficial effects on cardiac ischemia through reduction of premature ventricular contraction burden.

DETAILED DESCRIPTION:
Ischemic heart disease is a heterogeneous condition with multiple etiologies that may contribute to an imbalance in myocardial oxygen supply and demand, resulting in depletion of myocardial cellular energy stores. Management of this disease state is aimed primarily at improving myocardial oxygen supply through revascularization of underlying obstructive atherosclerosis, in conjunction with interventions to reduce myocardial oxygen demand. Chronic treatment is directed at reducing recurrent ischemic symptoms. Despite advances in anti-thrombotic therapy, coronary revascularization, and other preventive therapies, the risk of recurrent events in this population remains substantial, in particular among those patients with indicators of higher risk (e.g. ST-segment depression, or arrhythmias).

Ranolazine is a piperazine derivative that exerts anti-ischemic actions without a clinically significant effect on heart rate or blood pressure. At clinically relevant concentrations, ranolazine is an inhibitor of the slowly inactivating component of the cardiac sodium current (late INa), which may reduce the deleterious effects associated with the intracellular sodium and calcium overload that accompany and may promote myocardial ischemia. Ranolazine is available as an anti-anginal agent for patients with chronic angina. The Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST-Elevation Acute Coronary Syndromes (MERLIN)-TIMI 36 trial demonstrated the safety of ranolazine in patients after ACS and also showed it's anti-arrhythmic properties. In addition to the safety properties of ranolazine, the study showed that ranolazine had a significant anti-ischemic effect and patient's on therapeutic dosing.

In an analysis of the 6560 patients in MERLIN-TIMI 36, using a digital continuous electrocardiographic Holter monitor for ischemia (Lifecard CF, Delmar Reynolds was applied to patients at the time of randomization and remained in place for 7 days, including after hospital discharge). Findings showed that patients treated with ranolazine had significantly lower incidences of arrhythmias. Specifically, fewer patients had an episode of ventricular tachycardia lasting ≥8 beats, supraventricular tachycardia or new-onset atrial fibrillation. In addition, pauses ≥3 seconds were less frequent with ranolazine. Based on this report, further studies of the antiarrhythmic effects of ranolazine were warranted.

Premature ventricular complexes (PVCs) are a frequent occurrence in the presence of ischemic heart disease. A very high PVC burden can be symptomatic or occasionally result in a cardiomyopathy. The mechanism by which PVCs cause cardiomyopathies or symptoms is not well understood, but may be related to an increase in myocardial strain or demand. Reduction in PVC burden has been associated with both improvement in ejection fraction and symptoms. Ranolazine has also been shown to reduce PVC burden in patients already on optimal medical therapy. The estimate of the minimal number of PVCs required to be associated with a cardiomyopathy is around 10%. In fact, subjects that had evidence for PVCs on baseline 12 lead electrocardiogram were found to have a significantly higher risk of cardiovascular events.

Current strategies for managing complex cardiomyopathies driven by arrhythmias have been complicated by intolerance to medical therapy as well as the requirement for frequent titration and the development of tolerance. Patients with ischemic heart disease have limited options for antiarrhythmic medical therapy. Prior trials of flecainide and eicainide in patients with ischemic heart disease for control of ventricular arrhythmias resulted in a significant and deleterious proarrhythmic effect current options for management line on amiodarone which has significant liver, thyroid, and lung toxicities or sotalol which can have significant bronchospastic effects as well as QT prolongation or tedious and which has to be carefully dose in the setting of renal insufficiency to avoid significant QT prolongation and the risk for proarrhythmia.

While ICD therapy has been appropriate for patients with reduced ejection fraction and evidence for unstable ventricular arrhythmias/sudden cardiac death, frequent or low level ventricular arrhythmias such as nonsustained VT or frequent PVCs would not be treated by ICD therapy. Escalation of traditional nodal therapies such as beta blockers or calcium channel blockers is his often limited by marginal systolic blood pressures and/or symptoms.

With the increasing prevalence of ischemic heart disease, it is critically important to identify therapies that have a neutral response to heart rate and blood pressure, good safety profile, and can reduce ischemia and the burden ventricular arrhythmias. Ultimately, the hope is that they will reduce strain induced ischemic heart changes. To that end, investigation of the effects of ranolazine in patients with ischemic heart disease and an elevated burden of PVCs is of great interest.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years and older
* Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* History of ischemic heart disease (prior bypass or coronary stenting, documentation on cardiac catheterization, nuclear SPECT imaging, cardiac MR, stress echocardiography, or exercise stress testing). Subjects are not required to have chronic angina to be enrolled in the study
* Elevated PVC burden (1%) on prior Holter/event monitor in previous 12 months or evidence for PVC(s) on baseline ECG within prior 12 months.
* Sexually active females of childbearing potential must agree to utilize effective methods of contraception during heterosexual intercourse throughout the treatment period and for 14 days following discontinuation of the study medication

Exclusion Criteria:

* Hospitalization for hyperthyroidism, pericarditis, myocarditis, or pulmonary embolism within 4 weeks prior to screening
* Implantation of ICD or permanent pacemaker within 1 month of screening
* New York Heart Association (NYHA) Class III and IV heart failure or NYHA Class II heart failure with a recent decompensation requiring hospitalization or referral to a specialized heart failure clinic within 4 weeks prior to Screening.
* Myocardial infarction, unstable angina, or coronary artery bypass graft (CABG) surgery within three months prior to Screening or percutaneous coronary intervention (PCI) within 4 weeks prior to Screening
* Clinically significant valvular disease in the opinion of the Investigator
* Stroke within 1 months prior to Screening
* History of serious ventricular arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation) within 4 weeks prior to Screening
* Family history of long QT syndrome
* QTc ≥ 500 msec (Bazett) at Screening ECG if in sinus rhythm (SR). If in AF, evidence of QTc ≥ 500 msec (Bazett) within 4 weeks prior to Screening
* Prior heart transplant
* Cardiac ablation within 3 months prior to Screening, or planned ablation during the course of the study
* Need for concomitant treatment during the trial, with drugs or products that are strong inhibitors of CYP3A, or inducers of CYP3A. Such medications should be discontinued 5-half- lives prior to the Run-in period
* Use of grapefruit juice or Seville orange juice during the study
* Use of drugs that prolong the QT interval
* Previous use of ranolazine within 2 months prior to screening
* Prior use of ranolazine which was discontinued for safety or tolerability
* Use of dabigatran during the study
* Use of a greater than 1000 mg total daily dose of metformin during the study
* Hypokalemia (serum potassium < 3.5 mEq/L) at Screening that cannot be corrected to a level of potassium ≥ 3.5 mEq/L prior to randomization
* Moderate and severe hepatic impairment (ie, Child-Pugh Class B and C), abnormal liver function test defined as ALT, AST, or bilirubin > 2 x ULN at Screening
* Severe renal impairment defined as creatinine clearance ≤ 30 mL/min at Screening
* Females who are pregnant or are breastfeeding
* Exclusion of patients with Contraindications to use of RANEXA, including patients on CYP3A4 inducers/potent inhibitors, and patients with liver cirrhosis
* Exclusion of Patients with CrCl < 30 mL/min
* Limit dose of RANEXA to 500mg BID in patients on concurrent diltiazem/verapamil
* Limit concurrent simvastatin to 20 mg/day
* In the judgment of the Investigator, any clinically-significant ongoing medical condition that might jeopardize the subject's safety or interfere with the study, including participation in another clinical trial within the previous 30 days using a therapeutic modality which could have potential residual effects that might confound the results of this study
* Any technical issue (device related) which in the judgment of the investigator would disrupt adequate data collection or interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chester M Hedgepeth, MD, PhD, Principal Investigator — Brigham and Women's Cardiovascular Associates at Care New England
Locations (1):
- Kent Hospital, Warwick, Rhode Island, United States

REFERENCES:
- [Background] Scirica BM, Braunwald E, Belardinelli L, Hedgepeth CM, Spinar J, Wang W, Qin J, Karwatowska-Prokopczuk E, Verheugt FW, Morrow DA. Relationship between nonsustained ventricular tachycardia after non-ST-elevation acute coronary syndrome and sudden cardiac death: observations from the metabolic efficiency with ranolazine for less ischemia in non-ST-elevation acute coronary syndrome-thrombolysis in myocardial infarction 36 (MERLIN-TIMI 36) randomized controlled trial. Circulation. 2010 Aug 3;122(5):455-62. doi: 10.1161/CIRCULATIONAHA.110.937136. Epub 2010 Jul 19. PMID 20644019
- [Background] Scirica BM, Morrow DA, Budaj A, Dalby AJ, Mohanavelu S, Qin J, Aroesty J, Hedgepeth CM, Stone PH, Braunwald E. Ischemia detected on continuous electrocardiography after acute coronary syndrome: observations from the MERLIN-TIMI 36 (Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST-Elevation Acute Coronary Syndrome-Thrombolysis In Myocardial Infarction 36) trial. J Am Coll Cardiol. 2009 Apr 21;53(16):1411-21. doi: 10.1016/j.jacc.2008.12.053. PMID 19371824
- [Background] Kumar K, Nearing BD, Carvas M, Nascimento BC, Acar M, Belardinelli L, Verrier RL. Ranolazine exerts potent effects on atrial electrical properties and abbreviates atrial fibrillation duration in the intact porcine heart. J Cardiovasc Electrophysiol. 2009 Jul;20(7):796-802. doi: 10.1111/j.1540-8167.2009.01437.x. Epub 2009 Feb 27. PMID 19298570
- [Background] Scirica BM, Morrow DA, Hod H, Murphy SA, Belardinelli L, Hedgepeth CM, Molhoek P, Verheugt FW, Gersh BJ, McCabe CH, Braunwald E. Effect of ranolazine, an antianginal agent with novel electrophysiological properties, on the incidence of arrhythmias in patients with non ST-segment elevation acute coronary syndrome: results from the Metabolic Efficiency With Ranolazine for Less Ischemia in Non ST-Elevation Acute Coronary Syndrome Thrombolysis in Myocardial Infarction 36 (MERLIN-TIMI 36) randomized controlled trial. Circulation. 2007 Oct 9;116(15):1647-52. doi: 10.1161/CIRCULATIONAHA.107.724880. Epub 2007 Sep 5. PMID 17804441
- [Background] Kunadian B, Sutton AG, Vijayalakshmi K, Thornley AR, Gray JC, Grech ED, Hall JA, Harcombe AA, Wright RA, Smith RH, Murphy JJ, Shyam-Sundar A, Stewart MJ, Davies A, Linker NJ, de Belder MA. Early invasive versus conservative treatment in patients with failed fibrinolysis--no late survival benefit: the final analysis of the Middlesbrough Early Revascularisation to Limit Infarction (MERLIN) randomized trial. Am Heart J. 2007 May;153(5):763-71. doi: 10.1016/j.ahj.2007.02.021. PMID 17452151
- [Background] Ephrem G, Levine M, Friedmann P, Schweitzer P. The prognostic significance of frequency and morphology of premature ventricular complexes during ambulatory holter monitoring. Ann Noninvasive Electrocardiol. 2013 Mar;18(2):118-25. doi: 10.1111/anec.12010. Epub 2012 Nov 22. PMID 23530481
- [Background] Yokokawa M, Good E, Crawford T, Chugh A, Pelosi F Jr, Latchamsetty R, Jongnarangsin K, Armstrong W, Ghanbari H, Oral H, Morady F, Bogun F. Recovery from left ventricular dysfunction after ablation of frequent premature ventricular complexes. Heart Rhythm. 2013 Feb;10(2):172-5. doi: 10.1016/j.hrthm.2012.10.011. Epub 2012 Oct 23. PMID 23099051
- [Background] Ban JE, Park HC, Park JS, Nagamoto Y, Choi JI, Lim HE, Park SW, Kim YH. Electrocardiographic and electrophysiological characteristics of premature ventricular complexes associated with left ventricular dysfunction in patients without structural heart disease. Europace. 2013 May;15(5):735-41. doi: 10.1093/europace/eus371. Epub 2012 Nov 29. PMID 23194696
- [Background] Lee V, Hemingway H, Harb R, Crake T, Lambiase P. The prognostic significance of premature ventricular complexes in adults without clinically apparent heart disease: a meta-analysis and systematic review. Heart. 2012 Sep;98(17):1290-8. doi: 10.1136/heartjnl-2012-302005. Epub 2012 Jul 10. PMID 22781425
- [Background] Baman TS, Lange DC, Ilg KJ, Gupta SK, Liu TY, Alguire C, Armstrong W, Good E, Chugh A, Jongnarangsin K, Pelosi F Jr, Crawford T, Ebinger M, Oral H, Morady F, Bogun F. Relationship between burden of premature ventricular complexes and left ventricular function. Heart Rhythm. 2010 Jul;7(7):865-9. doi: 10.1016/j.hrthm.2010.03.036. Epub 2010 Mar 27. PMID 20348027
- [Background] Le VV, Mitiku T, Hadley D, Myers J, Froelicher VF. Rest premature ventricular contractions on routine ECG and prognosis in heart failure patients. Ann Noninvasive Electrocardiol. 2010 Jan;15(1):56-62. doi: 10.1111/j.1542-474X.2009.00340.x. PMID 20146783
- [Background] John RM, Tedrow UB, Koplan BA, Albert CM, Epstein LM, Sweeney MO, Miller AL, Michaud GF, Stevenson WG. Ventricular arrhythmias and sudden cardiac death. Lancet. 2012 Oct 27;380(9852):1520-9. doi: 10.1016/S0140-6736(12)61413-5. PMID 23101719
- [Background] Mountantonakis SE, Hutchinson MD. Indications for implantable cardioverter-defibrillator placement in ischemic cardiomyopathy and after myocardial infarction. Curr Heart Fail Rep. 2011 Dec;8(4):252-9. doi: 10.1007/s11897-011-0069-1. PMID 21769565
- [Background] Hickey KT, Reiffel J, Sciacca RR, Whang W, Biviano A, Baumeister M, Castillo C, Talathothi J, Garan H. Correlating perceived arrhythmia symptoms and quality of life in an older population with heart failure: a prospective, single centre, urban clinic study. J Clin Nurs. 2013 Feb;22(3-4):434-44. doi: 10.1111/j.1365-2702.2012.04307.x. PMID 23301579

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine
Started | 6
Completed | 2
Not Completed | 4
Not completed — Incomplete screening | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ranolazine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 78 [71 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Ranolazine on the PVC Burden Over 30 Days
Description: The change in percentage of PVC burden after taking Ranolazine 1000mg twice daily for 30 days
Time Frame: Baseline (7 day) Holter compared to day 30 (7 day) Holter
Population: The percentage of PVC's on Holter monitor at baseline compared to day 30 were used to determine the statistical significance of the data.
Measure: Mean (Full Range); unit: percentage of PVC burden
Arm/Group | Ranolazine
Number analyzed (Participants) | 2
percentage of PVC burden
  percentage of PVC burden at Baseline | 5.71 [5.52 to 9.73]
  percentage of PVC burden at Day 30 | 5.495 [1.2 to 9.73]

2. Primary Outcome: The Effect of Ranolazine on Cardiac Ischemia
Description: The effect of ranolazine on cardiac ischemia as measured by change in millimeters of ST segment deviation on ECG monitoring at Baseline and after 30 days of Ranolazine therapy (day 30).
Time Frame: Baseline and day 30
Measure: Mean (Full Range); unit: millimeters
Groups:
- Effect of Ranolazine on Cardiac Ischemia: Ranolazine 1000 mg tablet twice daily for 30 days
Arm/Group | Effect of Ranolazine on Cardiac Ischemia
Number analyzed (Participants) | 2
millimeters | 0 [0 to 0]

3. Secondary Outcome: Score on Seattle Angina Questionnaire at Baseline and at Day 30
Description: The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life). Angina symptoms may be felt as: chest pain, a heaviness, tightness or squeezing sensation in the chest, aching across the chest, particularly behind the breastbone. The pain may radiate to the neck, jaw, arms, back or teeth.
Time Frame: Baseline and day 30
Population: Score on Seattle Angina Questionnaire at Baseline and at day 30.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ranolazine
Number analyzed (Participants) | 2
score on a scale
  Baseline SAQ score for Angina Frequency | 95 [90 to 100]
  Day 30 SAQ score for Angina Frequency | 95 [90 to 100]
  Baseline score for Angina Stability | 50 [50 to 50]
  Day 30 SAQ score for Angina Stability | 50 [50 to 50]
  Baseline SAQ score for Physical Limitation | 94.445 [88.89 to 100]
  Day 30 SAQ score for Physical Limitation | 94.445 [88.89 to 100]
  Baseline SAQ score for Day 30 SAQ score Quality of | 79.165 [58.33 to 100]
  Day 30 SAQ score for Quality of Life | 87.5 [75 to 100]

4. Secondary Outcome: Number of Non-sustained Ventricular Tachycardia and Sustained Ventricular Arrhythmia Episodes on Holter Monitoring
Description: Number of non-sustained ventricular tachycardia episodes (>8 beats) and sustained ventricular arrhythmia episodes on Holter monitoring at baseline and at 30 days
Time Frame: Baseline and Day 30
Measure: Number; unit: number of episodes
Arm/Group | Ranolazine
Number analyzed (Participants) | 2
number of episodes
  Baseline Holter | 0
  Day 30 Holter | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ranolazine
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=6)
Syncopy (Cardiac disorders) | 1 (1) — Syncopy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT02360397/Prot_SAP_000.pdf